CLINICAL TRIAL: NCT00859105
Title: A Multicenter, Double-Blind, Vehical-Controlled Study Comparing Imiquimod Cream, 5% (Apotex Inc.) to Aldara™ Cream, 5%(3M Pharmaceutials, U.S.) and Aldara™ Cream, 5%(3M Pharmaceuticals, Canada) in the Treatments of Actinic Keratosis.
Brief Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Therapeutic Equivalence Study of Three Imiquimod Cream 5% Treatments for Patients With Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apotex Inc. (Industry)
Responsible Party: Bernice Tao, Director, Regulatory Affairs U.S.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMIQ-TOCR-01RB01-CE
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Imiquimod 5% (Experimental): Manufactured by Apotex
  Interventions: Drug: Imiquimod 5%: manufactured by Apotex
- Adara 5 % Cream US (Active Comparator): Manufactured by 3M, US.
  Interventions: Drug: Adara 5% Cream US
- Adara 5% Cream Canada (Active Comparator): Manufactured by 3M, Canada
  Interventions: Drug: Adara 5% Cream Canada
- Vehicle (Placebo Comparator): Manufactured by Apotex
  Interventions: Drug: Imiquimod Vehicle

INTERVENTIONS:
Drug: Imiquimod 5%: manufactured by Apotex — Treatment applied as a thin layer to target area once a day, 2 days each week, 16 weeks
  Arms: Imiquimod 5%
Drug: Adara 5% Cream US — Treatment applied as a thin layer to target area once a day, 2 days each week, for 16 weeks
  Arms: Adara 5 % Cream US
Drug: Adara 5% Cream Canada — Treatment applied as a thin layer to target area once a day, 2 days each week, for 16 weeks.
  Arms: Adara 5% Cream Canada
Drug: Imiquimod Vehicle — Treatment applied as a thin layer to target area once a day, 2 days each week, for 16 weeks
  Arms: Vehicle

SUMMARY:
Treatment, Randomized, Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor), Placebo Control, Parallel Assignment, Bio-equivalence Study

ELIGIBILITY:
Inclusion Criteria:

* Patients must have 4 to 8 clinically diagnosed, non-hyperkeratotic, non-hypertrophic AK lesions within a 25 cm2 contiguous treatment area on either the face or balding scalp
* Women either must be 1 year post-menopausal, surgically sterile, or agree to use a medically accepted form or birth control
* Free of any systemic or dermatological disorder
* Any skin type or race, providing the skin pigmentation will allow discernment of erythema

Exclusion Criteria:

* Basal cell or squamous cell carcinoma, or other possible confounding skin conditions (on face and scalp)
* History of cutaneous hyperreactivity or facial irritation to topical products
* Engaging in activities involving excessive or prolonged exposure to sunlight
* Receiving systemic cancer chemotherapy, psoralen plus UVA therapy, UVB therapy, laser abrasion, dermabrasion, glycolic acids, or chemical peels 6 months prior to study entry
* Currently using or have used systemic steroids 2 months prior to study
* Currently using or have used on the treatment area over-the-counter retinol products, corticosteroids, cryosurgery, curettage, 5-fluorouracil, or other topical actinic keratosis treatments 28 days prior to randomization
* Pregnant or nursing mothers
* History of allergy or sensitivity to imiquimod or related compounds or other components of the formulation
* Taking immunosuppressant medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary objectives are to establish the therapeutic equivalence of imiquimod cream 5%, manufactured by Apotex Inc. and two Aldara (imiquimod) creams, manufactured by 3M (US & Canada) , and to show superiority over vehicle in the treatment of AK. | 24 weeks

SECONDARY OUTCOMES:
The secondary objective is to compare the safety profiles of the three creams. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Brooks, Study Director — Apotex Inc.